CLINICAL TRIAL: NCT03457662
Title: Sonodynamic Therapy Manipulates Atherosclerosis Regression Trial on Patients With PAD and Claudication
Acronym: SMART-PAD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Ye Tian, Professor, MD, PhD, First Affiliated Hospital of Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ye Tian PAD
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Peripheral Arterial Disease; Atherosclerosis; Cardiovascular Diseases
MeSH Terms: conditions — Peripheral Arterial Disease; Atherosclerosis; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OMC and pseudo-SDT (Active Comparator): Optimal medical care (OMC) and pseudo-SDT are administrated in this arm. OMC is established according to the standards established by the 2016 ACC-AHA Guidelines for the Management of Patients with Peripheral Artery Disease in order to promote best practices for risk factor management.
  Interventions: Combination Product: OMC and pseudo-SDT
- OMC and SDT (Experimental): OMC and SDT are administrated in this arm.
  Interventions: Combination Product: OMC and SDT

INTERVENTIONS:
Combination Product: OMC and pseudo-SDT — OMC is established according to the 2016 ACC-AHA Guidelines for the Management of Patients with PAD. Pseudo-SDT combines saline injection and obstructed ultrasound exposure on targeted lesions to simulate real SDT progression.
  Arms: OMC and pseudo-SDT
Combination Product: OMC and SDT — OMC is established according to the 2016 ACC-AHA Guidelines for the Management of Patients with PAD. SDT treatment is the combination of sonosensitizer administration and target atherosclerotic lesions ultrasound exposure. Sinoporphyrin sodium (DVDMS) as sonosensitizer, is dissolved in 0.9% sodium solution for following skin test and intravenous injection. 0.01mg/ml DVDMS solution (0.1ml) is prepared for skin test followed by 0.04 mg/ml.DVDMS solution intravenous injection (0.2mg/kg). The target atherosclerotic lesions are marked on the corresponding skin with ultrasound guidance and underwent ultrasound exposure after 4 hours incubation. The therapeutic ultrasonic transducer is fixed to the marked skin site of each lesion.
  Arms: OMC and SDT

SUMMARY:
The purpose of this trial is to evaluate the safety and efficacy of sonodynamic therapy (SDT) on reducing atherosclerotic plaques inflammation among patients with symptomatic femoropopliteal peripheral artery disease.

DETAILED DESCRIPTION:
Atherosclerotic lower extremity PAD affects more than 202 million people in the worldwide. PAD is associated with a major decline in walking functional status and claudication is the most frequent symptom. Current claudication therapies are associated with significant limitations. Pharmacotherapy cilostazol and supervised exercise are recommended in 2016 AHA/ACC Guideline on the management of lower extremity PAD patients with claudication, but cilostazol may not achieve an ideal response rate, and supervised exercise efficacy may be limited by co-morbidities and medicare reimburse. Furthermore endovascular procedure may not be feasible, durable or cost-effective, especially in femoropopliteal arteries.

SDT is a novel anti-inflammatory regimen to atherosclerosis with non-invasive, plaque-based, macrophage-targeted characteristics. We hypothesize that reducing local arterial inflammation of affected limb will ameliorate claudication symptom in patients with PAD. The main objectives of this trial are to evaluate the efficacy and safety of SDT in patients with symptomatic femoropopliteal PAD.

Thirty-two eligible participants will be randomly assigned to SDT or sham-control groups. Results of PET/CT are the prespecified primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with atherosclerotic peripheral artery disease with symptoms of moderate to severe intermittent claudication (defined as ability to walk at least 2, but not more than 11 minutes on a graded treadmill test using the Gardner protocol)
* 2. Aged ≥40 years
* 3. Resting ABI < 0.9 or ABI decreases > 0.15 after treadmill test regardless of the ABI at rest
* 4. Presence of atherosclerotic plaque in femoropopliteal arteries including the common femoral artery, superficial femoral artery and popliteal artery as determined by: Duplex ultrasound imaging OR lower extremity computed Tomography Angiography (CTA) OR lower extremity magnetic resonance angiography (MRA) OR lower extremity catheter-based contrast arteriography. Each of these noninvasive and invasive anatomic assessments will identify patients with at least a 50% stenosis in the affected segment
* 5. Stable use of low to moderate dose statin and the permitted statin drugs/ doses: atorvastatin 20 mg, simvastatin 40 mg, rosuvastatin 10 mg, pravastatin, 40 mg, fluvastatin 80 mg or lovastatin 40 mg for at least 6 weeks prior to screening
* 6. Written informed consent

Exclusion Criteria:

* 1. Critical limb ischemia or other comorbid conditions that limit walking ability (claudication must be the consistent primary exercise limitation)
* 2. Inability to complete treadmill testing per protocol requirements
* 3. Two treadmill tests are completed at baseline to confirm reproducibility of results; those who deviates >25% are excluded
* 4. Severe aorto-iliac arteries stenosis or occlusion documented by noninvasive and invasive anatomic assessments
* 5. Active systemic inflammatory disease or have an infectious disease within 1 month prior to enrollment
* 6. Allergic to DVDMS
* 7. Diagnosis of porphyria
* 8. Pregnant women and nursing mothers
* 9. Contraindications of PET/CT
* 10. Concurrent enrollment in another clinical trial
* 11. Presence of any clinical condition that in the opinion of the principal investigator makes the patient not suitable to participate in the trial

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
Change in MDS TBR | Measured at baseline, 1month.
  The primary efficacy endpoint is the change of target-to-background ratio (TBR) within the most diseased segment (MDS) of index-leg artery at 30-day follow-up after treatment, defined as ratio of the standardized uptake value (SUV) in artery wall to background venous activity within the MDS of index- leg artery assessed by PET/CT.

SECONDARY OUTCOMES:
AS TBR change, (%) | Measured at baseline, 1month.
  Change from baseline to 30-day in active slice (AS) assessed by PET/CT. The mean max AS TBR is defined as average mean maximal TBR of only slices with TBR >1.6 from index-leg at baseline.
WV TBR change, (%) | Measured at baseline, 1month.
  Change from baseline to 30-day in whole vessel (WV) TBR assessed by PET/CT. The mean max WV TBR is defined as a single whole vessel average mean maximal TBR of all the slices that compose the index vessel.
PWT change, s | Measured at baseline, 1month.
  Change from baseline peak walking time (PWT) at 1 month is assessed by graded treadmill test (Gardner protocol). The patient continues the test until walking can no longer be tolerated because of claudication symptoms.
COT change, s | Measured at baseline, 1month.
  Change from baseline claudication onset time (COT) at 1 month is assessed by graded treadmill test (Gardner protocol). The patient continues the test until calf muscle discomfort is first noticed.
Pre-exercise ABI | Measured at baseline, 1month.
  Ankle-Brachial Index (ABI) is the ratio of the blood pressure at the ankle to the blood pressure of the upper arm. Pre- exercise ABI is collected routinely with the patient supine immediately prior to a treadmill test.
Diameter stenosis, (%) | Measured at baseline, 1month.
  Estimation of the maximum diameter stenosis of the affected segments by doppler ultrasound.
WIQ score | Measured at baseline, 1month.
  The Walking Impairment Questionnaire (WIQ) assesses the severity of the subjective walking impairment on distance, speed, and stair climbing scales. It is administered as a self report. Range: Minimum score is 0.2, maximum 100.
SF-36 score | Measured at baseline, 1month.
  The patient reported SF-36 data assesses subjective physical limitations, leg symptoms, social function, treatment satisfaction, and quality of life. It is administered as a self report. Higher scores are indicative of better outcome. The summary scores is compiled by taking the mean of five subscales generated from the original questions. Range: Minimum score is 11.1, maximum 85.

OTHER OUTCOMES:
The number and percentage of mildly/severely calcified sites | Measured at baseline, 1month.
  According to the Hounsfield unit calcium density of PET/CT, the arterial sites were divided into 3 groups: non-calcified sites (< 130 HU), mildly calcified sites (130-399 HU) and severely calcified sites (≥400 HU). The exploratory endpoints is the number and percentage of mildly/severely calcified sites.
The CT values of mildly and severely calcified sites | Measured at baseline, 1month.
  The exploratory endpoints is the CT values of mildly and severely calcified sites.
The TBR values of mildly and severely calcified sites | Measured at baseline, 1month.
  The exploratory endpoints is the TBR values of mildly and severely calcified sites.

CONTACTS AND LOCATIONS:
Overall Officials: YE TIAN, MD, PhD, Study Chair — First Affiliated Hospital of Harbin Medical University
Locations (1):
- The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

REFERENCES:
- [Derived] Jiang Y, Fan J, Li Y, Wu G, Wang Y, Yang J, Wang M, Cao Z, Li Q, Wang H, Zhang Z, Wang Y, Li B, Sun F, Zhang H, Zhang Z, Li K, Tian Y. Rapid reduction in plaque inflammation by sonodynamic therapy inpatients with symptomatic femoropopliteal peripheral artery disease:A randomized controlled trial. Int J Cardiol. 2021 Feb 15;325:132-139. doi: 10.1016/j.ijcard.2020.09.035. Epub 2020 Sep 20. PMID 32966832